CLINICAL TRIAL: NCT05214105
Title: Predicting Progression of Chronic Kidney Disease in Sickle Cell Anemia Using Machine Learning Models [PREMIER]
Brief Title: The Predictive Capacity of Machine Learning Models for Progressive Kidney Disease in Individuals With Sickle Cell Anemia
Acronym: PREMIER
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Tennessee (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); University of Illinois at Chicago (Other); University of Memphis (Other); University of North Carolina, Charlotte (Other); Wake Forest University (Other); University of North Carolina, Chapel Hill (Other)
Responsible Party: Principal Investigator, Kenneth Ataga MD, Principal Investigator, University of Tennessee
Other Study IDs: 2021-0746; 1R01HL159376-01 (NIH)
Record Dates: First submitted 2021-12-17; First posted 2022-01-28 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Sickle Cell Disease; Kidney Diseases, Chronic
Keywords: Machine Learning Models; Sickle Cell Disease; Chronic Kidney Disease; eGFR; Anemia, Sickle Cell; Albuminuria; Renal Insufficiency, Chronic; Renal Insufficiency; APOL1
MeSH Terms: conditions — Anemia, Sickle Cell; Renal Insufficiency, Chronic; Albuminuria; Renal Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Routine laboratory tests (CBC and chemistries), cystatin C, pregnancy tests (if female and of child-bearing capacity), urinalysis, spot urine albumin-creatinine ratio, and select plasma and urine biomarkers (ET-1, VEGF and soluble VCAM-1) and kidney function (urinary nephrin, KIM-1) and genomic DNA analyses for APOL1 G1/G2 alleles.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with sickle cell anemia: Prospective longitudinal study of patients with sickle cell anemia
  Interventions: Other: Biospecimen/DNA collection and analysis

INTERVENTIONS:
Other: Biospecimen/DNA collection and analysis — Patients will be followed longitudinally with collection of CBC and chemistries as well as research biomarkers (urine, plasma, and genomic materials).

SUMMARY:
This is a multicenter prospective, longitudinal cohort study which will evaluate the predictive capacity of machine learning (ML) models for progression of CKD in eligible patients for a minimum of 12 months and potentially for up to 4 years.

DETAILED DESCRIPTION:
Sickle cell disease (SCD) is characterized by a vasculopathy affecting multiple end organs, with complications including ischemic stroke, pulmonary hypertension, and chronic kidney disease (CKD). Albuminuria, an early measure of glomerular injury and a manifestation of CKD, is common in SCD and predicts progressive kidney disease. Kidney function decline is faster in SCD patients than in the general African American population. The prevalence of rapid decline, commonly defined as an estimated glomerular filtration rate (eGFR) decline of >3 mL/min/1.73 m2 per year, is ~ 31% in SCD, 3-fold higher than in the general population. Furthermore, high-risk Apolipoprotein 1 (APOL1) variants are associated with an increased risk of albuminuria and progression of CKD in SCD. It is well recognized that kidney disease, regardless of severity, is associated with increased mortality in SCD. The investigators have recently observed that rapid eGFR decline is also independently associated with increased mortality in SCD. Early identification of patients at risk for progression of CKD is important to address potentially modifiable risk factors, slow eGFR decline and reduce mortality.

The investigators have previously reported that machine learning (ML) models can identify patients at high risk for rapid decline in kidney function. In this study, the investigators propose the conduct of a prospective, multi-center study to build a ML-based predictive model for progression of CKD in adults with SCD. A model with high predictive capacity for progression of CKD not only affords risk-stratification, but also offers opportunities to modify known risk factors in hopes of attenuating kidney function loss and decreasing mortality risk.

The overall hypothesis is that ML models utilizing clinical and laboratory characteristics, additional biomarkers and genetic assessments have a higher predictive capacity for progression of CKD than persistent albuminuria alone in adults with sickle cell anemia.

ELIGIBILITY:
Inclusion Criteria:

1. HbSS or HbSβ0 thalassemia, 18 - 65 years old;
2. non-crisis, "steady state" with no acute pain episodes requiring medical contact in preceding 4 weeks;
3. ability to understand the study requirements.

Exclusion Criteria:

1. pregnant at enrollment;
2. poorly controlled hypertension;
3. long-standing diabetes with suspicion for diabetic nephropathy;
4. connective tissue disease such as systemic lupus erythematosus (SLE);
5. polycystic kidney disease or glomerular disease unrelated to SCD;
6. stem cell transplantation;
7. untreated human immunodeficiency virus (HIV), hepatitis B or C infection; h) history of cancer in last 5 years; i) End-stage renal disease (ESRD) on chronic dialysis; j) prior kidney transplantation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Four hundred patients with SCD (HbSS or HbSB0 thalassemia) between the ages of 18 and 65 who meet the eligibility criteria and provide consent to participate in the study, will be enrolled in this prospective longitudinal trial.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2022-07-05 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Develop two separate predictive models for progression of CKD (eGFR <90 mL/min/1·73 m2 and ≥25% drop in eGFR from baseline) and rapid eGFR decline (eGFR loss >3·0 mL/min/1·73 m2 per year) over the 12 months following the baseline clinic evaluation. | 12 months
  At each visit following the first 12 months, rate of eGFR change will be calculated using data from current and earlier visits.

SECONDARY OUTCOMES:
Alternate definitions of CKD progression as eGFR decline <90 mL/min/1·73 m2 and ≥50% drop in eGFR from baseline, and rapid eGFR decline as eGFR loss >5·0 mL/min/1·73 m2 per year will be evaluated. | 12 months
  At each visit following the first 12 months, rate of eGFR change will be calculated using data from current and earlier visits.
Evaluate the effect of APOL1 on the predictive capacity of ML models. Genomic DNA will be extracted from whole blood collected at baseline visits using standard techniques and genotyping will be performed as previously described. | 12 months
  At each visit following the first 12 months, rate of eGFR change will be calculated using data from current and earlier visits

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth I Ataga, MD, Principal Investigator — The University of Tennessee Health Science Center
Locations (3):
- United States (3):
  - University of Illinois at Chicago, Chicago, Illinois
  - Wake Forest University, Winston-Salem, North Carolina
  - The University of Tennessee Health Science Center, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be provided to other academic investigators, upon request, for the purposes of non-commercial research, utilizing institutional Material Transfer Agreement (MTA).
Supporting Information: Study Protocol, CSR, Analytic Code
Time Frame: From time of first patient enrollment to up to 7 years after completion of study.
Access Criteria: Requests for data from academic investigators will be approved by the Executive Committee of the PREMIER Study. Following approval, de-identified data will be shared in a secure manner.